CLINICAL TRIAL: NCT02972346
Title: Availability and Safety Study of ACTH to Treat Children SRNS/SDNS
Brief Title: Availability Study of ACTH to Treat Children SRNS/SDNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-044
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTH(+) (Experimental): routine treatment + ACTH
  Interventions: Drug: ACTH
- ACTH(-) (No Intervention): routine treatment

INTERVENTIONS:
Drug: ACTH — routine treatment plus ACTH 0.4 Unit/kg/day (Maximum 25Unit) for three consecutive days every 4 weeks
  Other Names: adrenocorticotropic hormone
  Arms: ACTH(+)

SUMMARY:
Primary nephrotic syndrome(NS) is a common children renal disease.About 20% primary nephrotic syndrome are steroid-dependent and steroid-resistant.Low serum cortisol is one of the main relapse reasons.Adrenocorticotropic hormone(ACTH)-induced steroidogenesis improve serum cortisol and also direct melanocortin receptors(MCRs) mediated protective effect on kidney cells. To investigate the efficacy and safety of ACTH to treat NS, total 42 children steroid resistant or steroid dependent NS is enrolling in this multicenter, prospective case series of prescription based treatment with ACTH for NS.

DETAILED DESCRIPTION:
Primary nephrotic syndrome(NS) is a common children renal disease.About 20% primary nephrotic syndrome are steroid-dependent and steroid-resistant.Low serum cortisol is one of the main relapse reasons.Adrenocorticotropic hormone(ACTH) can stimulates the adrenal cortex and its production of corticosteroids.ACTH also direct melanocortin receptors(MCRs) mediated protective effect on kidney cells. To investigate the efficacy and safety of ACTH to treat NS, total 42 children steroid resistant or steroid dependent NS is enrolling in this multicenter, prospective case series of prescription based treatment with ACTH for NS.

ELIGIBILITY:
Inclusion Criteria:

1. age:3-12 years old
2. primary nephrotic syndrome
3. SRNS or SDNS
4. Minor lesion or minimal change disease
5. Signed informed consent

Exclusion Criteria:

1. Second nephrotic syndrome
2. allergic to ACTH
3. Refuse to signed informed consent
4. have had ACTH treatment
5. serious complication

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
24-hour proteinuria excretion | 1.5 years

SECONDARY OUTCOMES:
times of relapse | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yufeng Li, Ph.D., Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526